CLINICAL TRIAL: NCT02039830
Title: Group Physiotherapy Compared to Individual Physiotherapy to Treat Urinary Incontinence in Aging Women: A Randomized Control Trial
Brief Title: Group Versus Individual Physiotherapy for Urinary Incontinence in Aging Women
Acronym: GROUP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Responsible Party: Principal Investigator, Chantal Dumoulin, Dr Chantal Dumoulin, researcher and laboratory director, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRC01:GROUP; CIHR258993 (Other Grant/Funding Number: Canadian Institute of Health Research)
Record Dates: First submitted 2013-12-12; First posted 2014-01-20 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Urinary Incontinence; Urinary Stress Incontinence
Keywords: female; aging; physiotherapy; pelvic floor; rehabilitation
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group physiotherapy (Experimental): 12 weekly treatment visit + daily home exercise program
  Interventions: Behavioral: Group physiotherapy
- Individual one-on-one physiotherapy (Active Comparator): 12 weekly treatment visit + daily home exercise program
  Interventions: Behavioral: Individual one-on-one physiotherapy

INTERVENTIONS:
Behavioral: Group physiotherapy — Multimodal Group physiotherapy 12 weeks of weekly Group physiotherapy treatments including education and pelvic floor muscle exercises
  Arms: Group physiotherapy
Behavioral: Individual one-on-one physiotherapy — Multimodal Individual physiotherapy 12 weeks of weekly Individual physiotherapy treatments including education and pelvic floor muscle exercises
  Arms: Individual one-on-one physiotherapy

SUMMARY:
The recommended treatment for urinary incontinence (UI) in women is individualised pelvic floor muscle (PFM) training, a costly and resource-intense approach; one Canada is currently unable to meet. This non-inferiority randomized control trial seeks to determine if group-based PFM training is as effective as individualised PFM training for treating UI in women 65 and over, and to establish the cost-effectiveness of both. Demonstrating that group-based treatment is at least as good as individualised one-on-one treatment and more cost-effective would warrant including group-based PFM training as a first-line UI treatment.

DETAILED DESCRIPTION:
The incidence of urinary incontinence (UI) in women increases with age but, unbeknownst to many, it is not a normal part of aging and, in most cases, can be effectively treated. Yet today, the majority of senior women go untreated due to a lack of both human and financial resources. In Canada, there are currently 3 million senior women. Over the next 15 years their numbers are expected to grow significantly, as will the incidence of UI. The number of senior women requiring treatment, let alone the future demand, makes it imperative that more cost-effective treatments be identified. The prevalence of UI in community- dwelling women 65 and over is high - 55% experience stress or urge UI, or even both, and of these, 20 to 25% are classified as having severe symptoms. Not only is UI a serious medical condition but it is also undeniably a social problem, engendering embarrassment and negative self-perceptions. It is associated with reduced social interactions and physical activities, with poor self-rated health, impaired emotional and psychological well-being and impaired sexual relationships. Moreover, it doubles women's risk of being admitted to a nursing home, independent of age or the presence of any other co-morbid conditions. It severely undermines a woman's right to healthy aging. Without doubt, this pervasive and serious condition requires immediate attention. Demographics, the negative impact on older women's functional autonomy and the current unmet treatment needs alone renders improving continence care for older women a priority for the Institute of Aging. This study aims to evaluate if group- based physiotherapy treatment is at least as good as individualized one-on-one physiotherapy treatment for treating urinary incontinence in aging women. The treatment efficacy will be assessed in 364 women (aged 60 years and older) suffering from stress or mixed urinary incontinence and recruited in 4 hospitals and in the community.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* suffering from stress urinary incontinence (SUI) or mixed urinary incontinence (MUI) symptoms
* at least 3 urinary incontinence episodes per week x 3 months or more
* ambulatory without the need of assisted device
* understand French or English instruction
* hormonal replacement stable for 6 months

Exclusion Criteria:

* present risk factors known to interfere with the effects of PFM training
* >2 degree Pop-Q
* body mass index >35
* chronic constipation
* have received physiotherapy or surgical treatment within the last year

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in the number of UI episodes | at recruitment, 13 weeks after recruitment and 12 months after recruitment, and 8 years after recruitment for those who completed the 12-month evaluation
  evaluated with a 7-day bladder diary

SECONDARY OUTCOMES:
Symptoms and degree to which UI-associated symptoms are troubling or bothersome | at recruitment, 13 weeks after recruitment and 12 months after recruitment, and 8 years after recruitment for those who completed the 12-month evaluation.
  evaluated using the International Consultation on Incontinence questionnaire on urinary incontinence (ICIQ-UI short form)
Symptoms and degree to which UI-associated symptoms are troubling or bothersome | at recruitment, 13 weeks after recruitment and 12 months after recruitment, and 8 years after recruitment for those who completed the 12-month evaluation.
  evaluated using the International Consultation on Incontinence questionnaire on nocturia (ICIQ-Nocturia)
Symptoms and degree to which UI-associated symptoms are troubling or bothersome | at recruitment, 13 weeks after recruitment and 12 months after recruitment.
  evaluated using the 24h PAD test
Symptoms and degree to which UI-associated symptoms are troubling or bothersome | at recruitment, 13 weeks after recruitment and 12 months after recruitment.
  evaluated using the International Consultation on Incontinence Questionnaire - Vaginal Symptoms Module (ICIQ-VS)
Symptoms and degree to which UI-associated symptoms are troubling or bothersome | at recruitment, 13 weeks after recruitment and 12 months after recruitment.
  evaluated using the International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS)
UI related QOL | at recruitment, 13 weeks after recruitment and 12 months after recruitment, and 8 years after recruitment for those who completed the 12-month evaluation
  evaluated using the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol)
UI related self-efficacy | at recruitment, 13 weeks after recruitment and 12 months after recruitment
  evaluated using the Geriatric self-efficacy index
UI related self-efficacy | 13 weeks after recruitment (recollection of what was before recruitment and what is now) and 12 months after recruitment, and 8 years after recruitment for those who completed the 12-month evaluation
  evaluated using the Broom PFM Self-efficacy scale
Costs related to interventions | at recruitment, 13 weeks after recruitment and 12 months after recruitment, and 8 years after recruitment for those who completed the 12-month evaluation
  evaluated using the modified Dowel-Bryant Incontinence Cost Index
Anthropometric measurements | at recruitment, 13 weeks after recruitment and 12 months after recruitment
  evaluated using height and weight measurements, which will be combined to report BMI in kg/m^2
PFM function | at recruitment, 13 weeks after recruitment and 12 months after recruitment
  evaluated combining digital palpation (Oxford scale), vaginal atrophy index and dynamometry
PFM morphology | at recruitment, 13 weeks after recruitment and 12 months after recruitment
  evaluated using transperineal US
Patient reported improvement and satisfaction | 13 weeks after recruitment and 12 months after recruitment
  evaluated using Patient global impression of improvement (PGI-I) and Benefit and willingness
Adherence to intervention and home exercises | after recruitment (once/week during 12 weeks), 13 weeks after after recruitment, 6 months after recruitment, at 9 months after recruitment, 12 months after recruitment, and 8 years after recruitment for those who completed the 12-month evaluation
  evaluated using homemade questionnaire including attendance to intervention and assiduity to home exercises program
Qualitative interview | 8 years after recruitement for those who completed the 12-month evaluation
  evaluated using homemade questionnaire including assiduity to lifestyle modification, changes in general health status, changes in medication, perceived change in UI symptoms, consultation with healthcare professionals for UI, and use of additional treatments for UI.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Dumoulin, Ph.D., Principal Investigator — Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Locations (1):
- Laboratoire incontinence et vieillissement CRIUGM, Montreal, Quebec, Canada

REFERENCES:
- [Background] Cacciari LP, Kouakou CR, Poder TG, Vale L, Morin M, Mayrand MH, Tousignant M, Dumoulin C. Group-based pelvic floor muscle training is a more cost-effective approach to treat urinary incontinence in older women: economic analysis of a randomised trial. J Physiother. 2022 Jul;68(3):191-196. doi: 10.1016/j.jphys.2022.06.001. Epub 2022 Jun 23. PMID 35753969
- [Background] Dumoulin C, Morin M, Danieli C, Cacciari L, Mayrand MH, Tousignant M, Abrahamowicz M; Urinary Incontinence and Aging Study Group. Group-Based vs Individual Pelvic Floor Muscle Training to Treat Urinary Incontinence in Older Women: A Randomized Clinical Trial. JAMA Intern Med. 2020 Oct 1;180(10):1284-1293. doi: 10.1001/jamainternmed.2020.2993. PMID 32744599
- [Background] Dumoulin C, Morin M, Mayrand MH, Tousignant M, Abrahamowicz M. Group physiotherapy compared to individual physiotherapy to treat urinary incontinence in aging women: study protocol for a randomized controlled trial. Trials. 2017 Nov 16;18(1):544. doi: 10.1186/s13063-017-2261-4. PMID 29145873
- [Derived] Cacciari LP, Morin M, Mayrand MH, Dumoulin C. Incontinence in Older Women: When to Expect Meaningful Leakage Reduction from Pelvic Floor Muscle Training. Int Urogynecol J. 2025 Dec 17. doi: 10.1007/s00192-025-06486-3. Online ahead of print. PMID 41405686
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322